CLINICAL TRIAL: NCT01100255
Title: Understanding the Glutamate System in Adults With Obsessive-Compulsive Disorder With N-methyl-D Aspartate Antagonist Ketamine
Brief Title: Pilot Study of Ketamine in Adults With Obsessive-Compulsive Disorder (OCD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 6906R/5883
Record Dates: First submitted 2010-04-05; First posted 2010-04-08 (Estimated); Results first posted 2016-10-27 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-01

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): 0.5mg/kg IV ketamine infusion over 40 minutes then IV saline infusion over 40 minutes
  Interventions: Drug: Ketamine infusion; Other: Saline
- Group B (Active Comparator): IV saline infusion over 40 minutes then 0.5mg/kg IV ketamine infusion over 40 minutes
  Interventions: Drug: Ketamine infusion; Other: Saline

INTERVENTIONS:
Drug: Ketamine infusion — 0.5mg/kg IV over 40 minutes
  Other Names: Ketamine hydrochloride
Other: Saline — saline infusion

SUMMARY:
In this study investigators are studying the effects of a drug called ketamine on the symptoms of Obsessive-compulsive disorder (OCD).

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) is a common psychiatric illness that affects up to 2-3% of the population. People with OCD experience anxiety-provoking, intrusive thoughts, known as obsessions, and feel compelled to perform repetitive behaviors, or compulsions. The only medications proven effective for OCD are serotonin reuptake inhibitors (SRIs), but even with SRI treatment, most patients continue to experience significant OCD symptoms, impaired functioning, and diminished quality of life. Recent evidence suggest that a different neurotransmitter, glutamate, may contribute to the symptoms in OCD. Medications that target glutamate hold promise for ameliorating symptoms for those patients continuing to suffer from OCD. In this study the investigators are recruiting patients to receive the drug ketamine, which is thought to modulate the neurotransmitter glutamate through the N-methyl-D-aspartate (NMDA), in a 2-week placebo controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55
* Physically healthy and not currently pregnant
* Primary Diagnosis of OCD
* Sufficient severity of symptoms
* Able to provide consent

Exclusion Criteria:

* Psychiatric conditions that make participation unsafe
* Currently on psychotropic medication
* Medical conditions that make participation unsafe
* Allergy to ketamine
* Any metal in the body

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2010-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn I. Rodriguez, M.D., Ph.D., Principal Investigator — Columbia-NYSPI-RFMH
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rodriguez CI, Kegeles LS, Flood P, Simpson HB. Rapid resolution of obsessions after an infusion of intravenous ketamine in a patient with treatment-resistant obsessive-compulsive disorder. J Clin Psychiatry. 2011 Apr;72(4):567-9. doi: 10.4088/JCP.10l06653. No abstract available. PMID 21527129
- [Result] Rodriguez CI, Kegeles LS, Levinson A, Feng T, Marcus SM, Vermes D, Flood P, Simpson HB. Randomized controlled crossover trial of ketamine in obsessive-compulsive disorder: proof-of-concept. Neuropsychopharmacology. 2013 Nov;38(12):2475-83. doi: 10.1038/npp.2013.150. Epub 2013 Jun 19. PMID 23783065
- [Result] Rodriguez CI, Kegeles LS, Levinson A, Ogden RT, Mao X, Milak MS, Vermes D, Xie S, Hunter L, Flood P, Moore H, Shungu DC, Simpson HB. In vivo effects of ketamine on glutamate-glutamine and gamma-aminobutyric acid in obsessive-compulsive disorder: Proof of concept. Psychiatry Res. 2015 Aug 30;233(2):141-7. doi: 10.1016/j.pscychresns.2015.06.001. Epub 2015 Jun 6. PMID 26104826

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A | Group B
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This was a cross over trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (10) | 32 (8) | 34 (9)
Gender [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Met and Exceeded Response Criteria of Yale-Brown Obsessive-Compulsive Scale.
Description: Patients given YBOCS (Yale Brown Obsessive-Compulsive Scale), a gold standard measure of obsessions and compulsions. For the YBOCS the minimum units are 0 and Maximum units on the total scale are 40. The higher the number on the YBOCS, the more severe the symptoms. Response was defined as at least a 35% reduction on the YBOCS.
Time Frame: 1 week
Measure: Number; unit: participants
Groups:
- Saline Infusion: IV saline infusion over 40 minutes
  Saline: saline infusion
- Ketamine Infusion: 0.5mg/kg IV infusion over 40 minutes
  Ketamine infusion: 0.5mg/kg IV over 40 minutes
Arm/Group | Saline Infusion | Ketamine Infusion
Number analyzed (Participants) | 15 | 15
participants | 0 | 5

ADVERSE EVENTS:
Groups:
- Saline Infusion: IV saline infusion over 40 minutes
- Ketamine Infusion: 0.5mg/kg IV ketamine infusion over 40 minutes
Arm/Group | Saline Infusion | Ketamine Infusion
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 4/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saline Infusion (N=15) | Ketamine Infusion (N=15)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3) — Dizziness resolved within 110min of the start of the infusion.
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) — Nausea resolved within 110min of the start of the infusion.
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) — Vomiting resolved within 110min of the start of the infusion.
Headache (Nervous system disorders) | 0 (0) | 2 (2) — Headache resolved within 110min of the start of the infusion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No